CLINICAL TRIAL: NCT06218953
Title: The Impact of Preoperative Anemia on Postoperative Anemia and Related Nutrient Abnormalities After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Yuntao Nie, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: CJBariatric004
Record Dates: First submitted 2023-12-25; First posted 2024-01-23 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Anemia; Bariatric Surgery
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the impact of preoperative anemia status on anemia and related nutrient abnormalities 1 year after bariatric surgery.

DETAILED DESCRIPTION:
This study aims to assess the impact of preoperative anemia status on anemia and related nutrient abnormalities (ferritin deficiency, vitamin B12 deficiency, folate deficiency, and low transferrin saturation level) at 1 year after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent bariatric surgery (sleeve gastrectomy and Roux-en-Y gastric bypass)
* Age between 16 and 70 years
* Patients who have complete 1-year follow-up data

Exclusion Criteria:

* Baseline renal failure
* Vegetarian
* Postoperative bleeding (it was defined as a drop in hemoglobin levels > 3 g/dL or a confirmed blood loss requiring treatment after surgery)

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent bariatric surgery aged between 16 and 70 years will receive follow-up for at least 1 year.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Odds ratio (OR) for anemia by preoperative anemia status | 1 year
  Multivariable logistic regression will be performed to assess the association between preoperative anemia and postoperative anemia. Several factors will be adjusted: sex, age, BMI, waist circumference, hip circumference, surgery, smoking, alcohol, hypertension, diabetes, hyperuricemia, hypercholesterolemia, and hypertriglyceridemia.

SECONDARY OUTCOMES:
Percentage of postoperative anemia | 1 year
  Percentage of postoperative anemia,, , and low transferrin saturation level.
Percentage of anemia severity | 1 year
  Percentage of anemia severity (mild: hemoglobin≥110g/L; moderate: hemoglobin≥80g/L; severe: hemoglobin<80g/L).
Percentage of ferritin deficiency | 1 year
  Percentage of ferritin deficiency, which is defined as ferritin less than 30 ng/mL.
Percentage of vitamin B12 deficiency | 1 year
  Percentage of ferritin deficiency, which is defined as vitamin B12 less than 150 pmol/L.
Percentage of folate deficiency | 1 year
  Percentage of folate deficiency, which is defined as folate less than 10 nmol/L.
Percentage of low transferrin saturation level | 1 year
  Percentage of low transferrin saturation level, which is defined as transferrin saturation less than 20%.

CONTACTS AND LOCATIONS:
Overall Officials: Yuntao Nie, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- Yuntao Nie, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Patient data must be obtained with the consent of the principal investigator.